CLINICAL TRIAL: NCT05326139
Title: The Effect of Topical Tranexamic Acid Application on Postoperative Periorbital Ecchymosis and Eyelid Edema in Rhinoplasty
Brief Title: Topical Tranexamic Acid Application in Rhinoplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ömer vural, Principal Investigator, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 25ovafbsi
Record Dates: First submitted 2022-04-02; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Ecchymosis; Eyelid; Edema; Rhinoplasty
Keywords: ecchymosis; rhinoplasty; edema; tranexamic acid
MeSH Terms: conditions — Ecchymosis; Edema | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Active Comparator): Group TA (n=25): TA ( Tranexamic acid, 250mg/2.5 ml inj ) soaked pledgets were placed under the skin flap to cover the osteotomy line
  Interventions: Drug: Tranexamic acid
- Isotonic saline (Placebo Comparator): Group Co (n=25): Isotonic saline ( NaCl, 0.9 %) soaked pledgets were placed under the skin flap to cover the osteotomy line
  Interventions: Other: Isotonic saline

INTERVENTIONS:
Drug: Tranexamic acid — TA-soaked pledgets were placed under the skin flap in such a way that both sides reach the osteotomy area and left for 5 minutes.
  Other Names: Transamin
  Arms: Tranexamic acid
Other: Isotonic saline — Isotonic saline -soaked pledgets were placed under the skin flap in such a way that both sides reach the osteotomy area and left for 5 minutes.
  Other Names: Mediflex %0.9 NaCl
  Arms: Isotonic saline

SUMMARY:
The aim of this study is to examine the effectiveness of topical Tranexamic acid application in overcoming periorbital ecchymosis and edema after rhinoplasty, which are common and do not have a standard treatment.

DETAILED DESCRIPTION:
All patients were informed individually about the procedures and written informed consent was obtained before the study. Patients who underwent rhinoplasty / septorhinoplasty operation between June 2021 and September 2021 with open technique were included in the study. Two groups with at least 25 individuals in each group were included in the study. Patients were appointed to either the control or TA group in a randomized-consecutive fashion. Patients younger than 18 years or older than 60 years, patients with a history of previous nasal operations, chronic medical conditions, hematologic disorders, fibrinolytic disorders and known allergy to tranexamic acid were excluded from the study. In group TA, TA-soaked pledgets were placed under the skin flap in such a way that both sides reach the osteotomy area and left for 5 minutes. In control group, isotonic saline-soaked pledgets were placed under the skin flap in the same way and left for 5 minutes. Surgical pledgets were prepared by nurse and given to the surgeon who did not know which group the pledget belonged to. Digital photographs were obtained by the surgeon who performed the operation on the first, third and seventh postoperative days. Eyelid edema and periorbital ecchymosis were scored via digital photographs separately by two expert surgeons at our institution independently using a graded scale ranging from 0 to 4. Digital photographs of the patients were shown to the examiners in alphabetical order, and information on which groups the patients belonged to was not given. The scores obtained from two different examiners were averaged. Statistical analyses were performed using IBM SPSS for Windows (IBM Corp., version 26.0, Armonk, NY, USA). The gender distribution of the groups was presented by number and percentage. Age, ecchymosis and edema degrees were presented by mean ± SD and median (minimum-maximum) values. The Chi-square test was used to compare the gender distribution of the groups. The patients' ecchymosis and edema scores were compared among groups using a Mann-Whitney U test. Comparisons within each group was evaluated with repeated measures analysis of variance test (Friedman test); if a difference was detected, the Wilcoxon signed rank test with Bonferroni correction was used to determine the group that made a difference. P ≤ .05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* primary open approach rhinoplasty under general anesthesia
* bilateral lateral osteotomies

Exclusion Criteria:

* Patients younger than 18 years
* Patients older than 60 years
* history of previous nasal operations
* chronic medical conditions,
* hematologic disorders
* known allergy to tranexamic acid

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Periorbital Ecchymosis | postoperative 1st day
  Ecchymosis around the eye as assessed using "4-point periorbital ecchymosis scale". Digital photographs were obtained on the first postoperative days. Periorbital ecchymosis were scored via digital photographs using a graded scale ranging from 0 to 4 point, higher scores mean a worse outcome.
Periorbital Ecchymosis | postoperative 3rd day
  Ecchymosis around the eye as assessed using "4-point periorbital ecchymosis scale". Digital photographs were obtained on the third postoperative days. Periorbital ecchymosis were scored via digital photographs using a graded scale ranging from 0 to 4 point, higher scores mean a worse outcome.
Periorbital Ecchymosis | postoperative 7th day
  Ecchymosis around the eye as assessed using "4-point periorbital ecchymosis scale". Digital photographs were obtained on the seventh postoperative days. Periorbital ecchymosis were scored via digital photographs using a graded scale ranging from 0 to 4 point, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Eyelid edema | postoperative 1st day
  Edema around the eye as assessed using "4-point eyelid edema scale". Digital photographs were obtained on the first postoperative days. Eyelid edema were scored via digital photographs using a graded scale ranging from 0 to 4 point, higher scores mean a worse outcome.
Eyelid edema | postoperative 3rd day
  Edema around the eye as assessed using "4-point eyelid edema scale". Digital photographs were obtained on the third postoperative days. Eyelid edema were scored via digital photographs using a graded scale ranging from 0 to 4 point, higher scores mean a worse outcome.
Eyelid edema | postoperative 7th day
  Edema around the eye as assessed using "4-point eyelid edema scale". Digital photographs were obtained on the seventh postoperative days. Eyelid edema were scored via digital photographs using a graded scale ranging from 0 to 4 point, higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: omer vural, Principal Investigator — Baskent University
Locations (1):
- Baskent University Faculty of Medicine, Çankaya, Ankata, Turkey (Türkiye)